CLINICAL TRIAL: NCT07377474
Title: A Study to Investigate the Safety and Effectiveness of the Technolas® TENEO 317 Model 2 Excimer Laser for Laser In Situ Keratomileusis (LASIK) Surgery to Treat Myopia or Myopic Astigmatism With Sphere Between 0.00D and -1.00D
Brief Title: A Study to Investigate the Safety and Effectiveness of the Technolas® TENEO 317 Model 2 Excimer Laser for Laser In Situ Keratomileusis (LASIK) Surgery to Treat Myopia or Myopic Astigmatism
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BL-SU01-TENLMY-6301
Record Dates: First submitted 2026-01-22; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Myopic Astigmatism
MeSH Terms: conditions — Astigmatism | interventions — Lasers, Excimer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- TENEO 317 Model 2 (1.28 US) Excimer Laser (Experimental)
  Interventions: Device: TENEO 317 Model 2 (1.28 US) Excimer Laser

INTERVENTIONS:
Device: TENEO 317 Model 2 (1.28 US) Excimer Laser — Surgery to Treat Myopia or Myopic Astigmatism with Sphere between 0.00D and -1.00D

SUMMARY:
This will be a multicenter, prospective, open label, non-randomized, single arm study evaluating the safety and effectiveness of the Technolas® TENEO 317 Model 2 (version 1.28 US software) Excimer Laser when used in LASIK surgery to treat myopia or myopic astigmatism. One or both eyes of a subject may be treated so long as both eyes meet all inclusion/exclusion requirements.

ELIGIBILITY:
Inclusion Criteria:

1. Are 22 years of age or older.
2. Have read, understood, and signed an ICF.
3. Have demonstrated stable refraction (i.e., a change of ≤ ± 0.5 D in sphere and cylinder) for a minimum of 12 months prior to surgery verified by consecutive refractions, medical records or prescription history.
4. Have myopic refractive error with or without astigmatism; sphere 0.00 D up to -1.00 D, cylinder between 0.00 D and -3.00 D; with a manifest refraction spherical equivalent (MRSE) between -.0375 D and -2.50 D.
5. Wears distance correction or has a need for distance correction.
6. Have manifest, distance best spectacle corrected visual acuity (BSCVA) of 20/25 (logMAR 0.1) or better in an operative eye.
7. Have equal to or less than 0.50 D spherical equivalent (SE) difference between cycloplegic and manifest refractions at Visit 1 (Pre-operative).
8. Have normal corneal topography as determined by the Investigator.
9. Anticipated postoperative stromal thickness of at least 350 microns.
10. Have discontinued use of contact lenses for at least 2 weeks (for hard or toric lenses) or 3 days (for soft contact lenses) prior to the pre-operative examination, and through the day of surgery.
11. All contact lens wearers must demonstrate a stable refraction (within ± 0.5 D), as determined by MRSE, on two consecutive examinations at least 1 week apart, in an eye to be treated and the axis of cylinder should not differ by more than 15 degrees from the baseline cycloplegic refraction.
12. Agree to emmetropia correction for each treated eye
13. Have the ability to lie flat without difficulty.
14. Are willing and able to comply with the schedule for all post-surgery follow-up visits.

Exclusion Criteria:

1. Subjects for whom the combination of their baseline corneal thickness and the planned operative parameters for the LASIK procedure would result in treatment depth less than 250 microns from corneal endothelium.
2. Acute or chronic disease or illness that would increase operative risk or confound the results of the study (e.g., dry eye, cataract, immuno-compromise, rheumatoid arthritis, clinically significant atopic disease, acne rosacea, autoimmune disease, endocrine disorders, lupus, systemic connective tissue disease, diabetes, or severe atopic disease).
3. Ocular conditions that may predispose the subject to future complications, including but not limited to:

   * History or evidence of retinal vascular disease
   * History or evidence of active corneal disease or infection (e.g., recurrent corneal erosion syndrome, herpes simplex or herpes zoster keratitis) in either eye.
   * History of or evidence of glaucoma or glaucoma suspect (e.g., IOP > 21 mmHg).
4. Eyes for which the baseline manifest subjective refraction exhibits a difference greater than 0.50 D in sphere power, or a difference greater than 0.50 D in cylinder power, or a difference in cylinder axis of more than 15 degrees compared to the baseline cycloplegic subjective refraction. For manifest cylinder of less than 0.50 D, the difference in cylinder axis will not be taken into consideration.
5. Subjects for whom the pre-operative assessment of the cornea indicates that one or both eyes are not suitable candidates for treatment based upon the Investigator's medical judgment.
6. Have evidence of retinal vascular disease.
7. Have a history of or have active corneal disease or infection (e.g., recurrent corneal erosion syndrome, herpes simplex or herpes zoster keratitis, etc.) in either eye.
8. Have a known sensitivity to any study medication.
9. Have central corneal scars affecting visual acuity or unstable keratometry with irregular mires in an eye considered for eligibility.
10. Presence of keratoconus, subclinical or forme fruste keratoconus, corneal dystrophy, unstable central keratometry readings with irregular mires, or other corneal irregularity (e.g., irregular astigmatism).
11. Had previous intraocular or corneal surgery in an eye considered for eligibility that might confound the outcome of the study or increase the risk to the subject.
12. Use chronic medications by any administration route that may increase risk to the subject or may confound the outcome of the study, including those known to affect wound healing (e.g., corticosteroids, antimetabolites, etc.).
13. Are taking medications contraindicated with LASIK such as isotretinoin (Accutane) or amiodarone hydrochloride (Cordarone).
14. Are known to be pregnant, lactating, or who plan to become pregnant during the course of the study.
15. Have known sensitivity to medications used for standard LASIK.
16. Have the presence of systemic disease likely to affect wound healing, e.g., autoimmune disease, systemic connective tissue disease, diabetes, or severe atopic disease.
17. Are participating in any other ophthalmic clinical trial within 30 days of screening or during this clinical trial.
18. Have an ocular muscle disorder including a strabismus or nystagmus, or other disorder affecting fixation.
19. Have a history of or evidence of glaucoma or are a glaucoma suspect.
20. Eyes with mesopic pupil size > 7.0 mm.
21. Have a Schirmer's pre-operative test without anesthesia < 4 mm/5 minutes

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
The percentage of eyes that achieve predictability (attempted versus achieved) of MRSE within ± 0.50 D | Assessed for approximately 12 months
The percentage of eyes that achieve predictability (attempted versus achieved) of MRSE within ± 1.00 D | Assessed for approximately 12 months
The percentage of eyes that achieve a UDVA of 20/40 or better | Assessed for approximately 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Rosangela Sonner, Study Director — Bausch & Lomb Incorporated

IPD SHARING:
Plan to Share IPD: No